CLINICAL TRIAL: NCT05039775
Title: Clitoral Therapy Device in Alleviating Sexual Dysfunction After Genital Mutilation of Females in Egypt.
Brief Title: Clitoral Therapy Device in Alleviating Sexual Dysfunction After Genital Mutilation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Hend Reda Sakr, Lecturer of Physical Therapy for Woman's Health, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hend3
Record Dates: First submitted 2021-09-01; First posted 2021-09-10 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Sexual Dysfunction; Sexual Arousal Disorder
Keywords: Sexual arousal disorder
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study group (Experimental): Forty married women, their ages will range from 20 to 45 years and all are suffering sexual dysfunction of sexual arousal and will use EROS-CTD Clitoral Therapy Device in addition to psychosexual support sessions and will be closely followed for three months.
  Interventions: Device: EROS device; Behavioral: Psychosexual support
- Control group (Other): Forty married women, their ages will range from 20 to 45 years and all are suffering sexual dysfunction of sexual arousal will receive psychosexual support sessions and will be closely followed after 3 months.
  Interventions: Behavioral: Psychosexual support

INTERVENTIONS:
Device: EROS device — Eros is a small, hand-held device fitted with a removable, replaceable small plastic cup used as a natural way to initiate female sexual response. It was originally cleared by the FDA in April 2000 for the treatment of Female Sexual Arousal Disorder (FSAD), which includes problems with sexual arousal and orgasm.
  Other Names: Clitoral therapy device
  Arms: Study group
Behavioral: Psychosexual support — Strategies are suggested to improve the couple's emotional connection and communication, when couples are being consulted, they are encouraged to focus on the strengths as well as weaknesses in their relationship. Homework assignments are given for the couple to practice skills, such as turning the idea of sexual obligation into pleasure, learning to focus on sensations rather than anxieties and communicating openly with their partner.
  Other Names: Psychosexual therapy

SUMMARY:
The aim of this study to determine the effect of clitoral therapy device EROS device/ on sexual dysfunction after genital mutilation.

DETAILED DESCRIPTION:
Little attention has been given to women who exposed to genital mutilation surgery in early age in the middle east. Most of them suffer from sexual dysfunction of sexual arousal and orgasm when they get in an intimate relation with their husbands after marriage. Clitoral therapy device may improve sexual arousal and alleviate sexual dysfunction symptoms to a great extent.

ELIGIBILITY:
Inclusion Criteria:

* All are suffering sexual dysfunction of sexual arousal and all referred from the family planning and reproductive health department, National research Center.

Exclusion Criteria:

* Metastatic disease, severe bowel or bladder sequelae, and significant comorbidities. Women with a history of sexual trauma or abuse, or undergoing current antidepressant therapy were excluded.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is targeting females who subjected to genital mutilation affecting their sexual life after marriage.
Enrollment: 80 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
The Female Sexual Function Index (FSFI). | Change from baseline sexual function at 3 months.
  Female sexual dysfunction has traditionally included disorders of desire. libido, arousal, pain/discomfort, and inhibited orgasm.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Abbassy, PhD, Principal Investigator — National Research Center
Locations (1):
- Badr University in Cairo, New Cairo, Badr City, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sakr HR, Ahmed YA, Kamel RM, Abdelhady RH, Elkalla RA, Georgui MA, Abd El-Khalek WO, El Ebrashy MH. Clitoral Therapy Device for Alleviating Sexual Dysfunction After Female Genital Mutilation: Randomized Controlled Trial. JMIR Rehabil Assist Technol. 2023 Apr 21;10:e43403. doi: 10.2196/43403. PMID 37083562